CLINICAL TRIAL: NCT01753219
Title: Effect of Suture for Mesh Fixation on Pain and Other Complications in Patients Undergoing Inguinal Hernia Repair: a Double-blind, Randomized Study Comparing the Lichtenstein With the Onstep Technique - the ONLI Trial.
Brief Title: Onstep Versus Lichtenstein, the Onli Trial.
Acronym: Onli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacob Rosenberg (Other)
Responsible Party: Sponsor-Investigator, Jacob Rosenberg, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Onli
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Hernia, Inguinal; Chronic Pain
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Onstep (Experimental): Participants in this group will have a inguinal hernia repair ad modum Onstep.
  Interventions: Procedure: Onstep
- Lichtenstein (Active Comparator): Participants in this group will receive a inguinal hernia repair ad modum Lichtenstein.
  Interventions: Procedure: Lichtenstein

INTERVENTIONS:
Procedure: Onstep
  Arms: Onstep
Procedure: Lichtenstein
  Arms: Lichtenstein

SUMMARY:
The objective of this study is to evaluate chronic pain and sexual dysfunction after inguinal hernia repair involving mesh fixation with sutures (Lichtenstein) compared with no mesh fixation (Onstep). The study hypothesis is that a smaller proportions of patients operated without mesh fixation (Onstep) will have chronic pain that impairs daily function.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnose of a primary groin hernia that requires surgical intervention.
* Eligible for procedure performed under general anesthesia

Exclusion Criteria:

* Not able to understand Danish, written and spoken.
* Emergency procedures
* Previous inguinal hernia on ipsilateral side.
* ASA score more than 3.
* Incarcerated or irreducible hernia.
* Local (site of surgery) or systemic infection.
* Contralateral hernia being operated at the same time or planned operated during follow-up.
* Other abdominal hernias being operated at the same time or planned operated during follow-up.
* Previous surgery that has impaired the sensation in the groin area.
* BMI > 40 or < 20.
* Daily intake of alcohol >5 units, 1 unit = 12g pure alcohol.
* Known disease that impairs central or peripheral nerve function.
* Concurrent malignant disease.
* Impairment of cognitive function (e.g. dementia).
* Chronic pain that requires daily medication.
* Mental disorder that requires medication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with chronic pain that impairs daily function | 6 month
  At the 6 month follow up, all participants will be asked to fill out questionnaires regarding pain. Questionnaire used will assess degree of pain and degree of impairment on daily function.
Proportion of patients with pain related impairment of sexual function | 6 month + 12 month
  At 6 and 12 month followup participants will be asked to fill out a questionnaire assessing pain related impairment of sexual function.
Proportion of patients with pain that impairs daily function | 12 month
  At the 12 month follow up, all pariticipants will be asked to fill out qestionnares regarding pain. Questionnaire used will assess degree of pain and degree of impairment of daily function.
Early postoperative pain | 10 days
  During the first 10 days, level of pain will be assessed using a Visual Analog Scale.

OTHER OUTCOMES:
30 day complications | 30 days
  Complications, occuring within the first 30 postoperative days will be recorded by telephone interview on day 30.
Cut to suture time | Peroperative
  The cut to suture time will be recorded by the staff in the operating room.
Lenght of hospital stay | Days
Time to return to normal daily activities | Days or weeks
Patients comfort | 6 and 12 month
  Patients comfort with the operated hernia be assessed using questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, Professor, Study Chair — University of Copenhagen, Herlev Hospital
Locations (4):
- Denmark (4):
  - Herlev Hospital, Herlev, Capital Region
  - Hospitalsenheden Horsens, Horsens, Region Midt
  - Hobro Sygehus, Hobro
  - Kolding Sygehus, Kolding

REFERENCES:
- [Background] Andresen K, Burcharth J, Rosenberg J. Lichtenstein versus Onstep for inguinal hernia repair: protocol for a double-blinded randomised trial. Dan Med J. 2013 Nov;60(11):A4729. PMID 24192245
- [Derived] Andresen K, Burcharth J, Fonnes S, Hupfeld L, Rothman JP, Deigaard S, Winther D, Errebo MB, Therkildsen R, Hauge D, Sorensen FS, Bjerg J, Rosenberg J. Sexual dysfunction after inguinal hernia repair with the Onstep versus Lichtenstein technique: A randomized clinical trial. Surgery. 2017 Jun;161(6):1690-1695. doi: 10.1016/j.surg.2016.12.030. Epub 2017 Mar 2. PMID 28262253
- [Derived] Andresen K, Burcharth J, Fonnes S, Hupfeld L, Rothman JP, Deigaard S, Winther D, Errebo MB, Therkildsen R, Hauge D, Sorensen FS, Bjerg J, Rosenberg J. Chronic pain after inguinal hernia repair with the ONSTEP versus the Lichtenstein technique, results of a double-blinded multicenter randomized clinical trial. Langenbecks Arch Surg. 2017 Mar;402(2):213-218. doi: 10.1007/s00423-016-1532-y. Epub 2016 Nov 11. PMID 27837273
- [Derived] Andresen K, Burcharth J, Fonnes S, Hupfeld L, Rothman JP, Deigaard S, Winther D, Errebo MB, Therkildsen R, Hauge D, Sorensen FS, Bjerg J, Rosenberg J. Short-term outcome after Onstep versus Lichtenstein technique for inguinal hernia repair: results from a randomized clinical trial. Hernia. 2015 Dec;19(6):871-7. doi: 10.1007/s10029-015-1428-8. Epub 2015 Oct 7. PMID 26445862